CLINICAL TRIAL: NCT02949830
Title: A Multicenter, Open-label Extension Study to Evaluate the Long-term Safety and Clinical Activity of Subcutaneously Administered ALN-AS1 in Patients With Acute Intermittent Porphyria Who Have Completed a Previous Clinical Study With ALN-AS1
Brief Title: A Study to Evaluate Long-term Safety and Clinical Activity of Givosiran (ALN-AS1) in Patient With Acute Intermittent Porphyria (AIP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-AS1-002; 2016-002638-54 (EudraCT Number)
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Intermittent Porphyria
Keywords: RNAi therapeutic; Porphyria; AIP; Heme/Haem Arginate
MeSH Terms: conditions — Porphyria, Acute Intermittent; Porphyrias | interventions — givosiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Givosiran (Experimental): At the beginning of this study, participants received either givosiran 2.5 mg/kg subcutaneous (SC) injection once monthly(QM), givosiran 5.0 mg/kg SC injection QM, or givosiran 5.0 mg/kg SC injection once every 3 months (Q3M). Within a year, all participants were transitioned to givosiran 2.5 mg/kg SC injection QM.
  Interventions: Drug: Givosiran

INTERVENTIONS:
Drug: Givosiran — Givosiran by subcutaneous (SC) injection.
  Other Names: ALN-AS1; Givlaari

SUMMARY:
The purpose of this study is to determine the long-term safety, tolerability and pharmacokinetics of givosiran (ALN-AS1) in AIP patients who completed study ALN-AS1-001 (NCT02452372).

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in Part C of study ALN-AS1-001 (NCT02452372)
* Not on a scheduled regimen of hemin
* Women of child bearing potential must have a negative serum pregnancy test, not be nursing, and use acceptable contraception
* Willing and able to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Clinically significant abnormal laboratory results
* Received an investigational agent (other than ALN-AS1) within 90 days before the first dose of study drug or are in follow-up of another clinical study
* History of multiple drug allergies or intolerance to subcutaneous injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (5):
- United States (3):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Galveston, Texas
- Clinical Trial Site, Stockholm, Sweden
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with acute intermittent porphyria (AIP) were enrolled at five sites in Sweden, United Kingdom and the United States.
Pre-assignment Details: Patients who completed parent study ALN-AS1-001 (NCT02452372) and met all eligibility criteria for this study (ALN-AS1-002) were enrolled.
Groups:
- Givosiran: At the beginning of this study, participants received either givosiran 2.5 mg/kg subcutaneous (SC) injection once monthly (QM), givosiran 5.0 mg/kg SC injection QM, or givosiran 5.0 mg/kg SC injection once every 3 months (Q3M). Within a year, all participants were transitioned to givosiran 2.5 mg/kg SC injection QM.
Period: Overall Study
Arm/Group | Givosiran
Started | 16
Completed | 14
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): All patients who received any amount of study drug.
Arm/Group | Givosiran
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 2
  White | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 15
  Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 6
  United Kingdom | 1
  United States of America | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Through Month 49
Population: SAS: All patients who received any amount of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Givosiran
Number analyzed (Participants) | 16
percentage of participants | 100

2. Secondary Outcome: The Pharmacodynamic (PD) Effect of Givosiran on Urine Levels of Delta-aminolevulinic Acid (ALA) as Measured by Percent Decrease From Baseline
Description: The PD effect of givosiran was evaluated by spot urine ALA levels normalized to spot urine creatinine levels.
Time Frame: Baseline; Month 48
Population: Patients from the PD Analysis Set (all patients who received any amount of study drug and who had at least 1 post-dose blood sample for PD), who were treated with givosiran 2.5 mg/kg SC injection QM. Values that occurred during a porphyria attack were excluded as a means of controlling for potential confounding by hemin. Overall number of participants analyzed is the number of participants available at the given time point.
Measure: Mean (Standard Error); unit: percent decrease
Arm/Group | Givosiran
Number analyzed (Participants) | 9
percent decrease | 92.531 (1.879)

3. Secondary Outcome: The Pharmacodynamic (PD) Effect of Givosiran on Urine Levels of Porphobilinogen (PBG) as Measured by Percent Decrease From Baseline
Description: The PD effect of givosiran was evaluated by spot urine PBG levels normalized to spot urine creatinine levels.
Time Frame: Baseline; Month 48
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percent decrease
Arm/Group | Givosiran
Number analyzed (Participants) | 9
percent decrease | 94.194 (2.617)

4. Secondary Outcome: Annualized Rate of Composite Porphyria Attacks
Description: Porphyria attacks were defined as meeting all of the following criteria: an acute episode of neurovisceral pain in the abdomen, back, chest, extremities and/or limbs, no other medically determined cause, and required treatment with intravenous (IV) dextrose or hemin, carbohydrates, or analgesics, or other medications such as antiemetics at a dose or frequency beyond the participant's usual daily porphyria management. Composite porphyria attacks included porphyria attacks that required hospitalization, urgent healthcare visit, or intravenous (IV) hemin administration at home. The annualized attack rate (AAR) was calculated as the number of composite porphyria attacks/total person-years.
Time Frame: Through Month 48
Population: SAS: All patients who received any amount of study drug.
Measure: Number; unit: composite attacks/total person-years
Arm/Group | Givosiran
Number analyzed (Participants) | 16
composite attacks/total person-years | 0.4

5. Secondary Outcome: Annualized Rate of Hemin Administration
Description: The annualized rate of hemin administration was evaluated by annualized days of hemin use, which is calculated as the number of doses of hemin administered/total person-years.
Time Frame: Through Month 49
Population: SAS: All patients who received any amount of study drug.
Measure: Number; unit: hemin doses/total person-years
Arm/Group | Givosiran
Number analyzed (Participants) | 16
hemin doses/total person-years | 0.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) are any AE with onset after the first administration of study drug through the end of exposure, or any event that was present at Baseline but worsened in severity or was subsequently considered drug-related by the Investigator (up to approximately 52 months).
Arm/Group | Givosiran
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Givosiran (N=16)
Abdominal pain (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sinusitis bacterial (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Givosiran (N=16)
Neutrophilia (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 1
Teething (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Discomfort (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 7
Feeling abnormal (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site discolouration (General disorders) | 2
Injection site dryness (General disorders) | 1
Injection site erythema (General disorders) | 6
Injection site indentation (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site pruritus (General disorders) | 4
Injection site rash (General disorders) | 2
Injection site swelling (General disorders) | 2
Injection site urticaria (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 2
Allergy to animal (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Oral allergy syndrome (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 8
Pharyngitis streptococcal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 2
Varicella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Venomous sting (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Albumin urine present (Investigations) | 1
Anticoagulation drug level below therapeutic (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Bilirubin conjugated increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood homocysteine increased (Investigations) | 1
Blood sodium decreased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
Carbon dioxide increased (Investigations) | 1
Coronavirus test positive (Investigations) | 1
Creatinine urine increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 3
Glomerular filtration rate decreased (Investigations) | 3
International normalised ratio increased (Investigations) | 4
Lipase increased (Investigations) | 4
Liver function test increased (Investigations) | 1
Protein urine present (Investigations) | 1
Prothrombin level increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine ketone body present (Investigations) | 1
Urine output decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Gluten sensitivity (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Panic attack (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 3
Menorrhagia (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 1
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Superficial vein prominence (Vascular disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is intended that after completion of the study, the data are to be submitted for publication in a scientific journal and/or for reporting at a scientific meeting. A copy of any proposed manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission, and according to any additional publication details in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT02949830/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT02949830/SAP_001.pdf